CLINICAL TRIAL: NCT04990440
Title: A Phase 2a, Multicenter, Randomized, Placebo-Controlled, Double-Blind, Interventional Study to Assess the Efficacy, Safety, Pharmacokinetics, and Immunogenicity of Multiple IV Doses of Bermekimab for the Treatment of Adult Participants With Moderate-to-Severe Atopic Dermatitis
Brief Title: A Study of Bermekimab for the Treatment of Adult Participants With Moderate-to-Severe Atopic Dermatitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Premature study termination (efficacy)
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CR109057; 2020-005900-21 (EudraCT Number); 77474462ADM2003 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-07-27; First posted 2021-08-04 (Actual); Results first posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-04

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic | interventions — bermekimab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A: Bermekimab Dose 1 (Experimental): Participants will receive bermekimab Dose 1 or placebo as an intravenous (IV) infusion weekly from Week 0 to Week 15.
  Interventions: Drug: Bermekimab; Drug: Placebo
- Part B: Bermekimab Dose 2 (Experimental): Participants will receive bermekimab Dose 2 or placebo as an IV infusion weekly from Week 0 to Week 15.
  Interventions: Drug: Bermekimab; Drug: Placebo
- Part C: Bermekimab Dose 3 (Experimental): Participants will receive bermekimab or placebo at a higher or lower dose (not less than [<] Dose 1) than Part B, but with a maximum dose of Dose 3 IV weekly based on pharmacokinetic (PK), pharmacodynamic (PD), efficacy, and safety analysis.
  Interventions: Drug: Bermekimab; Drug: Placebo

INTERVENTIONS:
Drug: Bermekimab — Participants will receive bermekimab IV.
  Other Names: JNJ-77474462
Drug: Placebo — Participants will receive placebo IV.

SUMMARY:
The purpose of this study is to evaluate the efficacy of Bermekimab, compared with placebo, in participants with moderate-to-severe atopic dermatitis (AD).

ELIGIBILITY:
Inclusion Criteria:

* Have atopic dermatitis (AD) for at least 1 year (365 days) prior to the first administration of study intervention as determined by the investigator through participant interview and/or review of the medical history
* Have a history of inadequate response to treatment for AD with topical medications or for whom topical treatments are otherwise medically inadvisable (example, due to important side effects or safety risks)
* Have an Eczema Area and Severity Index (EASI) score greater than or equal to (>=) 16 at screening and at baseline
* Must sign an informed consent form (ICF) indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study
* Must be willing to undergo 4 skin biopsies
* Have an Investigator Global Assessment (IGA) score >=3 at screening and at baseline
* Have an involved body surface area (BSA) >=10 percent (%) at screening and at baseline

Exclusion Criteria:

* Has a current diagnosis or signs or symptoms of severe, progressive, or uncontrolled renal, cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances
* Has ever received any Human interleukin-1 (IL-1) antagonist (example, including but not limited to anakinra, rilonacept)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2022-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (11):
- United States (6):
  - Dawes Fretzin Clinical Research Group, Indianapolis, Indiana
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Vital Prospects Clinical Research Institute, PC, Tulsa, Oklahoma
  - Modern Research Associates, Dallas, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
- Argentina (5):
  - CARE - Centro de Alergia y Enfermedades Respiratorias, Buenos Aires
  - Conexa Investigacion Clinica S.A., CABA
  - STAT Research S.A., CABA
  - Clínica Adventista Belgrano, CABA
  - CINME - Centro de Investigaciones Metabolicas, Ciudad de Buenos Aires

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 9 participants were screened, of which, only 6 participants were enrolled and randomized.
  Planned Part C was not performed due to premature study termination.
Groups:
- Part A: Placebo: Participants received placebo matching to bermekimab as an intravenous (IV) infusion weekly from Week 0 through Week 6.
- Part A: Bermekimab 800 mg IV: Participants received bermekimab 800 milligrams (mg) as an IV infusion weekly from Week 0 through Week 6.
- Part B: Bermekimab 1200 mg IV: Participants received bermekimab 1200 mg as an IV infusion weekly from Week 0 through Week 6.
Period: Overall Study
Arm/Group | Part A: Placebo | Part A: Bermekimab 800 mg IV | Part B: Bermekimab 1200 mg IV
Started | 1 | 4 | 1
Completed | 1 | 4 | 0
Not Completed | 0 | 0 | 1
Not completed — Sponsor's Decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Placebo | Part A: Bermekimab 800 mg IV | Part B: Bermekimab 1200 mg IV | Total
Number analyzed (Participants) | 1 | 4 | 1 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 19 | 34.5 (16.34) | 47 | 34 (15.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 0 | 3
  Male | 1 | 1 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 1 | 3 | 0 | 4
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  ARGENTINA | 1 | 3 | 0 | 4
  UNITED STATES | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Eczema Area and Severity Index (EASI)-75 (Greater Than or Equal to [>=] 75 Percent [%] Improvement From Baseline)
Description: Percentage of participants with EASI-75 (>=75% improvement from Baseline in EASI score) was planned to be reported in this outcome measure. The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema (E), infiltration (I), excoriation (Ex) and lichenification (L) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. The severity of the clinical signs of AD for each of 4 body regions was scored on a 4-point scale: 0=absent, 1=mild, 2=moderate and 3=severe. The area of AD involvement on each of the 4 anatomic regions was assessed as a percentage by body area: 0=no eruption, 1=1% to 9%, 2=10% to 29%, 3=30% to 49%, 4=50% to 60%, 5=70% to 80% and 6=90% to 100%. The total score is the sum of the four body-region scores ranged from 0.0 to 72.0, with higher scores reflecting greater disease severity.
Time Frame: Week 16
Population: The full analysis set (FAS) included all participants who were randomized at Week 0 and received at least 1 dose of study intervention. Due to premature study termination, planned data collection and analysis could not be performed for this outcome measure.
Arm/Group | Part A: Placebo | Part A: Bermekimab 800 mg IV | Part B: Bermekimab 1200 mg IV
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Serum Concentrations of Bermekimab Over Time
Description: Serum concentrations of bermekimab was planned to be reported up to Week 20 but due to premature study termination, planned data collection and analysis could not be performed for this outcome measure.
Time Frame: Up to Week 20
Population: Pharmacokinetic (PK) analysis set included all participants who received at least one dose of bermekimab and had at least one post-dose sample collection.
Arm/Group | Part A: Placebo | Part A: Bermekimab 800 mg IV | Part B: Bermekimab 1200 mg IV
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With Antibodies to Bermekimab (Anti-Drug Antibodies [ADAs] and Neutralizing Antibodies [NAbs])
Description: Number of participants with ADAs and NAbs to bermekimab was planned to be reported up to Week 16 but due to premature study termination, planned data collection and analysis could not be performed for this outcome measure.
Time Frame: Up to Week 16
Population: Immunogenicity analysis set included all participants who received at least one dose of bermekimab and had at least one post-dose sample collection.
Arm/Group | Part A: Placebo | Part A: Bermekimab 800 mg IV | Part B: Bermekimab 1200 mg IV
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. Any AE occurring at or after the initial administration of study intervention up to end of study was considered as treatment-emergent. Due to premature study termination, data collected up to Week 6 were analyzed and reported for this outcome measure.
Time Frame: Up to Week 6
Population: The safety analysis set included all participants who received at least 1 dose of study intervention and were analyzed based on the treatment they actually received regardless of the treatment groups to which they were assigned.
Measure: Number; unit: Percentage of participants
Arm/Group | Part A: Placebo | Part A: Bermekimab 800 mg IV | Part B: Bermekimab 1200 mg IV
Number analyzed (Participants) | 1 | 4 | 1
Percentage of participants | 100 | 75 | 100

5. Secondary Outcome: Percentage of Participants With Treatment-emergent Serious Adverse Events (TESAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse event (SAE) was any untoward medical occurrence that at any dose resulted in death, was life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a suspected transmission of any infectious agent via a medicinal product. Any SAEs occurring at or after the initial administration of study intervention up to end of the study was considered as treatment-emergent. Due to premature study termination, data collected up to Week 6 were analyzed and reported for this outcome measure.
Time Frame: Up to Week 6
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Part A: Placebo | Part A: Bermekimab 800 mg IV | Part B: Bermekimab 1200 mg IV
Number analyzed (Participants) | 1 | 4 | 1
Percentage of participants | 0 | 0 | 100

6. Secondary Outcome: Percentage of Participants With AEs Leading to Discontinuation of Study Intervention
Description: Percentage of participants with AEs leading to discontinuation of study intervention was reported. An AE was any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. Due to premature study termination, data collected up to Week 6 were analyzed and reported for this outcome measure.
Time Frame: Up to Week 6
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Part A: Placebo | Part A: Bermekimab 800 mg IV | Part B: Bermekimab 1200 mg IV
Number analyzed (Participants) | 1 | 4 | 1
Percentage of participants | 0 | 0 | 0

7. Secondary Outcome: Percentage of Participants With AEs Reasonably Related to Study Intervention
Description: Percentage of participants with AEs reasonably related to study intervention was reported. An AE was any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. Due to premature study termination, data collected up to Week 6 were analyzed and reported for this outcome measure.
Time Frame: Up to Week 6
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Part A: Placebo | Part A: Bermekimab 800 mg IV | Part B: Bermekimab 1200 mg IV
Number analyzed (Participants) | 1 | 4 | 1
Percentage of participants | 0 | 25 | 0

8. Secondary Outcome: Percentage of Participants With Adverse Events of Infusion-related Reactions
Description: Percentage of participants with adverse events of infusion-related reactions was reported. An AE was any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. Due to premature study termination, data collected up to Week 6 were analyzed and reported for this outcome measure.
Time Frame: Up to Week 6
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Part A: Placebo | Part A: Bermekimab 800 mg IV | Part B: Bermekimab 1200 mg IV
Number analyzed (Participants) | 1 | 4 | 1
Percentage of participants | 0 | 25 | 0

9. Secondary Outcome: Percentage of Participants With AEs of Infections
Description: Percentage of participants with AEs of infections (including serious infections and infections requiring oral or parenteral antimicrobial treatment) was reported. An AE was any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. Due to premature study termination, data collected up to Week 6 were analyzed and reported for this outcome measure.
Time Frame: Up to Week 6
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Part A: Placebo | Part A: Bermekimab 800 mg IV | Part B: Bermekimab 1200 mg IV
Number analyzed (Participants) | 1 | 4 | 1
Percentage of participants | 0 | 50 | 0

10. Secondary Outcome: Percentage of Participants With Clinically Significant Abnormalities in Vital Signs
Description: In this outcome measure, percentage of participants with clinically significant abnormalities in vital sign (respiratory rate) was reported. The clinical significance was determined by the investigator. Due to premature study termination, data collected up to Week 6 were analyzed and reported for this outcome measure.
Time Frame: Up to Week 6
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Part A: Placebo | Part A: Bermekimab 800 mg IV | Part B: Bermekimab 1200 mg IV
Number analyzed (Participants) | 1 | 4 | 1
Percentage of participants | 100 | 0 | 0

11. Secondary Outcome: Percentage of Participants With Clinically Significant Abnormalities in Laboratory Tests
Description: In this outcome measure, percentage of participants with >=2 National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) grade in laboratory parameter 'clinical chemistry-potassium (normal range: 3.5 to 5.2 mmol/L)' was reported. Grading was done as: Grade 1 (=mild), Grade 2 (=moderate), Grade 3 (=severe) and Grade 4 (=potentially life-threatening). The clinical significance was determined by the investigator. Due to premature study termination, data collected up to Week 6 were analyzed and reported for this outcome measure.
Time Frame: Up to Week 6
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Part A: Placebo | Part A: Bermekimab 800 mg IV | Part B: Bermekimab 1200 mg IV
Number analyzed (Participants) | 1 | 4 | 1
Percentage of participants | 0 | 25 | 0

12. Secondary Outcome: Percentage of Participants With Both Validated Investigator Global Assessment for Atopic Dermatitis (vIGA-AD) Score of 0 or 1 and a Reduction From Baseline of >=2 Points
Description: Percentage of participants with both vIGA-AD score of 0 or 1 and a reduction from baseline of >=2 points was reported. IGA was an assessment scale used to determine severity of AD and clinical response to treatment on a 5-point scale ranged from 0 to 4, where 0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe. Higher scores indicated greater severity. The IGA score was selected using the morphological descriptors that best described the overall appearance (erythema and population/infiltration) of the AD lesions at a given time point.
Time Frame: Week 16
Population: FAS included all participants who were randomized at Week 0 and received at least 1 dose of study intervention. Due to premature study termination, planned data collection and analysis could not be performed for this outcome measure.
Arm/Group | Part A: Placebo | Part A: Bermekimab 800 mg IV | Part B: Bermekimab 1200 mg IV
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Percentage of Participants With Improvement (Reduction) of Eczema-related Itch Numeric Rating Scale (NRS) Score of >=4 From Baseline Among Participants With a Baseline Itch Value >=4
Description: Percentage of participants with improvement (reduction) of eczema-related itch NRS score of >=4 from baseline among participants with a baseline itch value >=4 was reported in this outcome measure. The eczema skin pain and itch NRS was a 2-item (pain and itch) patient-reported outcome (PRO) developed by the sponsor that participants used to rate the severity of their eczema-related skin pain and itch daily. To rate the severity of eczema-related itch, participants were asked the following question: 'how would you rate your itch at the worst moment during the previous 24 hours' and the response was scored on a scale of 0 (no itch) to 10 (worst itch imaginable).
Time Frame: Week 16
Population: as for outcome 12
Arm/Group | Part A: Placebo | Part A: Bermekimab 800 mg IV | Part B: Bermekimab 1200 mg IV
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: Percentage of Participants With EASI-90
Description: Percentage of participants with EASI-90 was planned to be reported. The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema (E), infiltration (I), excoriation (Ex) and lichenification (L) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. The severity of the clinical signs of AD for each of 4 body regions was scored on a 4-point scale: 0=absent, 1=mild, 2=moderate and 3=severe. The area of AD involvement on each of the 4 anatomic regions was assessed as a percentage by body area: 0=no eruption, 1=1% to 9%, 2=10% to 29%, 3=30% to 49%, 4=50% to 60%, 5=70% to 80% and 6=90% to 100%. The total score is the sum of the four body-region scores ranged from 0.0 to 72.0, with higher scores reflecting greater disease severity.
Time Frame: Week 16
Population: as for outcome 12
Arm/Group | Part A: Placebo | Part A: Bermekimab 800 mg IV | Part B: Bermekimab 1200 mg IV
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Week 6
Description: The safety analysis set included all participants who received at least 1 dose of study intervention and were analyzed based on the treatment they actually received regardless of the treatment groups to which they were assigned. Due to premature study termination, adverse events data collected up to Week 6 were analyzed and reported in this section.
Arm/Group | Part A: Placebo | Part A: Bermekimab 800 mg IV | Part B: Bermekimab 1200 mg IV
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/4 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/4 | 1/1
Other Adverse Events (participants affected / at risk) | 1/1 | 3/4 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Placebo (N=1) | Part A: Bermekimab 800 mg IV (N=4) | Part B: Bermekimab 1200 mg IV (N=1)
Accidental Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Placebo (N=1) | Part A: Bermekimab 800 mg IV (N=4) | Part B: Bermekimab 1200 mg IV (N=1)
Otitis Externa (Infections and infestations) | 0 | 1 | 0
Vulvovaginal Candidiasis (Infections and infestations) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 1 | 2 | 0

LIMITATIONS AND CAVEATS:
The study 77474462ADM2001 (NCT04791319) was terminated due to futility analysis and no dose-response was observed. Based on study 77474462ADM2001 result, the current study (77474462ADM2003) was terminated early and thereby the planned Part C was not performed. Due to premature study termination, data collected up to Week 6 were analyzed and reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2021-11-23): https://cdn.clinicaltrials.gov/large-docs/40/NCT04990440/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-24): https://cdn.clinicaltrials.gov/large-docs/40/NCT04990440/SAP_001.pdf